CLINICAL TRIAL: NCT07389135
Title: The Role of Heart Rate Variability and Anxiety in Predicting Emergence Agitation in Patients Undergoing Septorhinoplasty : A Prospective Observational Study
Brief Title: Heart Rate Variability and Anxiety as Predictors of Emergence Agitation After Septorhinoplasty
Status: Not yet recruiting | Type: Observational
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Mahmut Sami TUTAR, Associate Professor, Department of Anesthesiology and Reanimation, Konya City Hospital
Other Study IDs: 26.06.2025/ 737-737-10
Record Dates: First submitted 2026-01-20; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Emergence Agitation; Heart Rate Variability (HRV); Septorhinoplasty
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Emergence Agitation: Participants who exhibit emergence agitation during early recovery in the PACU, defined as a Richmond Agitation-Sedation Scale (RASS) score ≥ +1 within the first 30 minutes after arrival to the PACU.
- No Emergence Agitation: Participants who do not exhibit emergence agitation during early recovery in the PACU, defined as RASS < +1 throughout the first 30 minutes after arrival to the PACU.

SUMMARY:
This prospective observational study aims to evaluate whether preoperative heart rate variability (HRV) and anxiety are associated with, and can help predict, emergence agitation in adult patients undergoing elective septorhinoplasty under general anesthesia. Preoperative anxiety will be assessed using a visual analog scale (VAS) and the State-Trait Anxiety Inventory (STAI-1). Resting HRV will be recorded preoperatively using a chest-strap heart rate monitor and HRV metrics (e.g., SDNN, RMSSD, LF/HF) will be derived. Emergence agitation will be assessed in the post-anesthesia care unit (PACU) using the Richmond Agitation-Sedation Scale (RASS) during the early recovery period. Secondary observations will include early postoperative events such as postoperative nausea and vomiting (PONV) and laryngospasm. The study is planned to enroll approximately 100 participants.

DETAILED DESCRIPTION:
Emergence agitation is a clinically relevant phenomenon during early recovery from general anesthesia and may be influenced by individual autonomic function and psychological factors. Heart rate variability (HRV) reflects autonomic nervous system activity, while preoperative anxiety has been associated with adverse recovery profiles in some surgical settings. This study will investigate the relationship between preoperative HRV, anxiety, and emergence agitation in adults undergoing elective septorhinoplasty.

This is a single-center, prospective observational study. Eligible patients will be adults scheduled for elective septorhinoplasty under routine general anesthesia care. Before surgery, participants will complete a preoperative anxiety assessment using a visual analog scale (VAS) and the State-Trait Anxiety Inventory (STAI-1). Resting HRV will be recorded preoperatively while the patient is at rest using a chest-strap heart rate monitor; time- and frequency-domain parameters (e.g., SDNN, RMSSD, LF/HF) will be calculated.

Postoperatively, emergence agitation will be evaluated in the PACU using the Richmond Agitation-Sedation Scale (RASS) at regular intervals during the first 30 minutes of recovery; emergence agitation will be defined as a RASS score ≥ +1. Additional peri-recovery observations will include postoperative nausea and vomiting (PONV) assessed over the first 24 hours and the occurrence of laryngospasm based on clinical criteria. The primary objective is to determine whether preoperative HRV metrics and anxiety measures are associated with emergence agitation and to explore their predictive value.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years
* ASA physical status I-II
* Scheduled for elective septorhinoplasty under general anesthesia
* Able to provide informed consent and complete questionnaires

Exclusion Criteria:

* ASA physical status III or higher
* Pregnancy or breastfeeding
* Known dysrhythmia/arrhythmia or autonomic dysfunction, or use of medications that may affect autonomic function/HRV
* Diagnosed anxiety disorder
* Use of preoperative anxiolytic medication
* Inability to understand/complete the anxiety scales/questionnaires
* Emergency surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (18-65 years, ASA I-II) undergoing elective septorhinoplasty under routine general anesthesia at a single center.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Emergence Agitation | First 30 minutes after arrival to the PACU
  Emergence agitation will be assessed in the post-anesthesia care unit (PACU) using the Richmond Agitation-Sedation Scale (RASS). EA will be defined as a RASS score ≥ +1 at any assessment during the observation period.

SECONDARY OUTCOMES:
Incidence of Laryngospasm | From extubation until discharge from the PACU
  Occurrence of clinically diagnosed laryngospasm during emergence from anesthesia or early recovery.
Postoperative Nausea and Vomiting (PONV) | Within 24 hours postoperatively
  Incidence and severity of postoperative nausea and vomiting assessed using a 4-point scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to institutional policies and data privacy concerns.